CLINICAL TRIAL: NCT00349999
Title: Protective Immunity to Human Cholera in Bangladesh-EGD Substudy
Brief Title: Protective Immunity to Human Cholera in Bangladesh
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0103; 5U01AI058935-14 (NIH)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2009-10

CONDITIONS: Cholera
Keywords: Vibrio cholerae, Cholera, Bangladesh, esophagogastroduodenoscopy, sub-study
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Duodenal biopsy samples and blood.

GROUPS / COHORTS (1):
- 1: 18 males and non pregnant females, ages 18-45, with acute cholera.

SUMMARY:
The purpose of this study is to better understand how the body fights and protects against cholera. Two hundered fifty people presenting to the International Centre for Diarrhoeal Diseases Research, Bangladesh, admitted with acute cholera, 50 of whom (healthy, nonpregnant, 18-45 year olds) will be enrolled in this substudy of mucosal immunity involving duodenal biopsy. The remainder of the study is observational, involving collection of stool, vomit, and blood samples only. The biopsy requires a flexible tube with a camera be inserted through the mouth into the stomach and intestine. During this procedure, small samples will be collected from the intestine. The study includes medical history, physical, blood testing, hospitalization and urine pregnancy testing. This study will last for 5 years and patients will participate for 3 years.

DETAILED DESCRIPTION:
Diarrheal diseases are some of the most common causes of morbidity and mortality in the world today. Unfortunately, effective vaccines for most of the infectious causes of diarrhea are not yet available. Vibrio cholerae (V cholerae) is an important infectious cause of severe secretory diarrhea in humans. The purpose of this study is to assess the duration of immune responses in a group of 250 individuals, aged 2-60 years, presenting to the International Centre for Diarrheal Diseases Research, Bangladesh (ICDDR,B) hospital who are admitted with acute cholera. Fifty of these participants will be enrolled in a substudy of mucosal immunity involving duodenal biopsy. This protocol focuses exclusively on the subset of 50 study participants (healthy 18-45 year old non pregnant subjects) enrolled in the substudy of mucosal immunity involving duodenal biopsy. This study is linked to DMID protocol 06-0045. The remainder of the study is observational, involving collection of stool, vomit, and blood samples only (DMID protocol 06-0045). A duodenal biopsy will be performed on enrollment or the next day and at Day 30. Twenty five subjects will undergo a third duodenal biopsy after 6 months of follow-up and 25 subjects will undergo a third duodenal biopsy after 12 months follow-up. The objectives of this study are as follows: to measure immune responses directed against Vibrio cholerae antigens and evaluate the development of anti-V cholerae memory B cells in study participants with cholera; to assess the duration of the immune responses following an episode of cholera; and to correlate the duration of antigen-specific, antibody-secreting cells for various cholera antigens in duodenal tissue with measurements of the duration of immunity based on antibody responses in serum, as well as circulating antigen-specific memory B cells. This is a single site study with a 5 year duration requiring three years of patient participation.

ELIGIBILITY:
Inclusion Criteria:

For the esophagogastroduodenoscopy (EGD) substudy of 50 study participants

* Admission to the International Centre for Diarrhoeal Diseases Research, Bangladesh (ICDDR,B) with acute cholera
* Male or nonpregnant female [pregnancy will be excluded by urine human chorionic gonadotropin (HCG) testing]
* Age 18 to 45 years, inclusive
* Residence in Dhaka city
* Provision of informed consent for enrollment in study
* Expressed interest and availability to fulfill the study requirements

Exclusion Criteria:

For the esophagogastroduodenoscopy (EGD) substudy of 50 study participants

* Participation in any other investigational drug, device or vaccine trial at present or within the past 30 days
* Known allergy to midazolam or topical anesthetics
* Presence of comorbid conditions, including:
* heart disease
* pulmonary disease
* liver disease
* kidney disease
* bleeding disorder
* neurologic disorder
* an additional intestinal disorder
* pregnancy
* anemia (hemoglobin < 12 g/dl for males or < 11 g/dl for female)
* hypotension (systolic blood pressure less than or equal to 85 mm Hg or diastolic blood pressure less than or equal to 55 mm Hg, measured in the supine position once just prior to procedure)
* hypertension (systolic blood pressure greater than or equal to 150 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg, measured in the supine position once just prior to procedure)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18 males and nonpregnant females, without comorbid conditions, ranging from 18 to 45 years of age, inclusive, who are admitted to the International Centre for Diarrhoeal Research, Bangladesh (ICDDR,B) with acute cholera.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Serum antibody responses to V cholerae Lipopolysaccharide (LPS) and Cholera Toxin, B Subunit (CTB) (and other antigens as needed) on Days 2, 7, and 30 and at Months 3, 6, 9, 12, 18, 24, 30, and 36 following enrollment. | Days 2, 7, and 30 and at Months 3, 6, 9, 12, 18, 24, 30, and 36 following enrollment.
Mucosal responses to V cholerae LPS and CTB (and other antigens as needed) on Days 2 and 30 (in 50 study participants) and at Month 6 (25 study participants) and Month 12 (25 study participants) following enrollment. | Days 2 and 30 (in 50 participants) and at Month 6 (25 study participants) and Month 12 (25 study participants) following enrollment.
Memory B and T cell responses to V cholerae LPS and CTB (and other antigens as needed) on Days 2 and 30 and at Months 3, 6, 9, 12, 18, 24, 39, and 36 following enrollment. | Days 2 and 30 and at Months 3, 6, 9, 12, 18, 24, 39, and 36 following enrollment..

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Hospital - International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh